CLINICAL TRIAL: NCT04048187
Title: Quality Control of CE-Certified Phonak Hearing Aids - 2019_23
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PMCF data, originally planned to be collected withthis study, are collected using another methodology
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Sonova2019_23
Record Dates: First submitted 2019-08-06; First posted 2019-08-07 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phone Application (Experimental)
  Interventions: Device: Phone Application

INTERVENTIONS:
Device: Phone Application — Phone application is developed to adjust hearing aids. It incorporates functionalities like volume control and program change.

SUMMARY:
Phonak Hearing Devices pass through different development and study phases. At an early stage, feasibiltiy studies are conducted to investigate new algorithms, features and functions in an isolated manner. If the benefit is proven, their performance is then investigated regarding interpendency between all available algorithms, features and functions running in parallel in a hearing aid (pivotal/pre-validation studies) and, resulting from the pre-validation studies, they get optimized. Prior to product launch, the Phonak Hearing Systems get reviewed by a final quality control in terms of clinical trials. This is a pre-validation study, investigating improved algorithms, features, functions and wearing comfort. This will be a clinical investigation which will be conducted mono centric at Sonova AG Headquarters based in Stäfa (Switzerland).

DETAILED DESCRIPTION:
This study will prove the overall performance and system context of the functionality in the mobile application in combination with hearing devices under real life conditions with experienced hearing aid users. The enduser should be able to adjust their hearing aid settings by App.

The app allows the user to change e.g. the loudness of the hearing aids and to create hearing scenarios by themselves. The users also shall be able to accept a conferecene call, which they will receive from the investigator via App.

This will be a clinical investigation which will be conducted mono centric at Sonova AG Headquarters based in Stäfa (Switzerland).

ELIGIBILITY:
Inclusion Criteria:

* experienced hearing aid users (minimum age: 18 years, moderate to moderate/severe hearing loss)
* modern subjects with an affinity to new technology
* willingness and interest in testing Apps
* owning a compatible smartphone
* Healthy outer ear
* willingness to wear behind the ear hearing aids
* Informed Consent as documented by signature

Exclusion Criteria:

* the audiogramm is not in the fitting range of the intended hearing aid
* limited mobility and not in the position to attend weekly appointments in Stäfa (Switzerland)
* participant is not able to describe experiences and hearing impressions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-09-06 (Actual)

PRIMARY OUTCOMES:
Successful creation of a Custom Sceario (%) | 4 weeks
  Endusers of the phoneApp are able to add a custum scenario to the app.
Successful answering of conference call (%) | 2 weeks
  Endusers of the phoneApp are able to answering the conference call?

CONTACTS AND LOCATIONS:
Locations (1):
- Sonova AG, Stäfa, Switzerland